CLINICAL TRIAL: NCT03302624
Title: A Study on the Follow-up of Long-term Renal Function After Acute Kidney Injury in ICU
Brief Title: Follow-up of Long-term Renal Function After Acute Kidney Injury in ICU
Acronym: SURIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-351
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Acute Kidney Injuries; Quality of Life; Chronic Kidney Disease; Renal Replacement Therapy
Keywords: acute kidney injury; quality of life; Renal replacement therapy; Intensive care unit
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who were included in ELVIS study

SUMMARY:
Acute kidney injury (AKI) involves poor prognosis in ICU patients. The renal prognosis at long term is unknown.

The study will determine chronic kidney injury incidence and quality of life, five years after AK during ICU stay.

DETAILED DESCRIPTION:
Prospective study. All patients who participated ELVIS study (clinical trials: 00875069) can be enrolled in SURIA.

Patients are contacted by telephone. Investigator delivery objective and honest information. If patients accepts the study, answers will be collected.

Collected data are: creatinine serum, two surveys (quality of life and activities of daily living), date of onset of renal replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

ICU Patients included in ELVIS study, AKI requiring renal replacement therapy Length of ICU stay ≥ 48h

Exclusion Criteria:

Pregnant or nursing woman's job

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 506 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of chronic kidney disease | 5 years after the first acute kidney injury requiring renal replacement therapy
  incidence of chronic kidney disease in patients who had an acute kidney injury during their ICU stay and requiring an renal replacement therapy

SECONDARY OUTCOMES:
severity of CKD according to the International Classification of Chronic Kidney Disease | 5 years after the first acute kidney injury requiring renal replacement therapy
  Kidney function will be measured by creatinine serum or chronic dialysis or kidney transplantation
impact of the renal replacement therapy on long-term renal function | 5 years after the first acute kidney injury requiring renal replacement therapy
  Intermittent or continuous renal replacement therapy. Data collected in the database from ELVIS study. Kidney function will be measured by creatinine serum or chronic dialysis
quality of life | 5 years after the first acute kidney injury requiring renal replacement therapy
  Quality of life will be assessed with the Q5D score
Activities of daily living | 5 years after the first acute kidney injury requiring renal replacement therapy
  Activities of daily living will be assessed with the Katz adjustment scales
Mortality | 5 years after the first acute kidney injury requiring renal replacement therapy
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre LAUTRETTE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Soum E, Timsit JF, Ruckly S, Gruson D, Canet E, Klouche K, Argaud L, Garrouste-Orgeas M, Mariat C, Vincent F, Cayot S, Darmon M, Bohe J, Schwebel C, Bouadma L, Dupuis C, Souweine B, Lautrette A. Predictive factors for severe long-term chronic kidney disease after acute kidney injury requiring renal replacement therapy in critically ill patients: an ancillary study of the ELVIS randomized controlled trial. Crit Care. 2022 Nov 29;26(1):367. doi: 10.1186/s13054-022-04233-4. PMID 36447221